CLINICAL TRIAL: NCT04263090
Title: A Phase1/2a Study of Rigosertib Plus Nivolumab in Stage IV Lung Adenocarcinoma Patients With KRAS Mutation Who Progressed on First-Line Treatment
Brief Title: Rigosertib Plus Nivolumab for KRAS+ NSCLC Patients Who Progressed on First-Line Treatment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Bristol-Myers Squibb (Industry); Traws Pharma, Inc. (Industry)
Responsible Party: Principal Investigator, Rajwanth Veluswamy, Assistant Professor, Hematology & Medical Oncology, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GCO 19-2243
Record Dates: First submitted 2020-02-05; First posted 2020-02-10 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Non-small Cell Lung Cancer; Adenocarcinoma; Stage IV
Keywords: KRAS; Metastatic; Rigosertib; Immunotherapy; Nivolumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Adenocarcinoma; Neoplasm Metastasis | interventions — ON 01910; Nivolumab

STUDY DESIGN:
Intervention Model Description: Dose-escalating Phase I study followed by a Phase 2a dose-expansion phase.
  Rigosertib escalation will occur with three dose levels: Dose D1: 280mg twice daily, Dose D2: 560mg qAM, 280mg qPM, Dose D3: 560mg twice daily. Nivolumab will be dosed at the standard fixed dose of 240mg.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rigosertib + Nivolumab (Experimental): Rigosertib + Nivolumab in metastatic KRAS+ lung adenocarcinoma patients
  Interventions: Drug: Rigosertib; Drug: Nivolumab

INTERVENTIONS:
Drug: Rigosertib — Rigosertib will be dosed twice a day for 21 consecutive days, followed by 7 days off treatment (each cycle duration: 28 days). Rigosertib escalation will occur with three dose levels (dose D1: 280mg twice daily; dose D2: 560mg qAM, 280mg qPM; dose D3: 560mg twice daily).
Drug: Nivolumab — Nivolumab will be dosed once ever 2 weeks (twice per 28-day cycle; standard fixed dose of 240mg).

SUMMARY:
A Phase1/2a Study of Rigosertib plus Nivolumab in Stage IV Lung Adenocarcinoma Patients with KRAS Mutation who Progressed on First-Line Treatment

DETAILED DESCRIPTION:
This is an open-label, dose-escalating Phase I study followed by a Phase 2a dose-expansion phase to study the combination of Rigosertib and Nivolumab in metastatic Kirsten rat sarcoma positive (KRAS+) lung adenocarcinoma patients who have progressed on standard first line treatment. Study patients will have satisfied the inclusion/exclusion criteria enumerated in this protocol. The Phase I dose escalation plan will start with an accelerated titration design (ATD) using single patient cohorts until grade 2 toxicity is experienced. At that point, the ATD will be terminated and the dose escalation will enter a standard 3+3 design based on dose-limiting toxicities (DLT). The MTD (Phase 1 primary endpoint) is defined as the highest dose for which at most 1 patient out of 6 experiences a DLT.

Rigosertib escalation will occur with three dose levels (dose D1: 280mg twice daily; dose D2: 560mg in the morning (qAM), 280mg in the evening (qPM); dose D3: 560mg twice daily; taken by mouth for 21 consecutive days of the 28 day cycle), based on previous dose escalation studies in other malignancies, while Nivolumab dose will be fixed at the standard dose (240mg every 2 weeks, given intravenously).

Once the MTD is determined, an additional planned 12 patients will be enrolled in the expansion phase to further study toxicity and to determine preliminary efficacy endpoints including ORR (phase 2a primary endpoint), PFS, and OS (secondary endpoints) of the combination.

ELIGIBILITY:
Inclusion criteria

* Be willing and able to provide written informed consent for the trial.
* Be at least 18 years of age on the day of signing informed consent.
* Have a histologically or cytologically confirmed diagnosis of Stage IV metastatic lung adenocarcinoma (AJCC version 8) with mutation analysis by next generation sequencing (NGS) confirming KRAS mutation either at time of diagnosis or at progression on first line treatment.
* Have progressed on or intolerant of standard of care first-line treatment with anti-programmed death-ligand 1 (PD1) checkpoint inhibitor monotherapy or anti-PD1 checkpoint inhibitor in combination with platinum doublet chemotherapy for Stage IV metastatic lung adenocarcinoma. The last cycle of first-line treatment must occur at least 28 days prior to administration of trial drugs (i.e., washout period)
* Have measurable disease per RECIST 1.1 as assessed by the local site investigator/radiology. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesion.
* Have a life expectancy of at least 3 months.
* Have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2.
* Have adequate organ function as indicated by the following laboratory values in Table 1. Specimens must be collected within 14 days prior to the start of trial.
* Patient must be willing and able to provide blood samples (12 green tops tubes, roughly 100mL) at the time points indicated in the Study Calendar.
* Patient must be willing and able to have core needle biopsies (Goal 4-8 biopsies, final number to be determined by the surgeon and radiologist performing the procedure as safe) of tumor prior to initiation of study drug, and at time points indicated in the Study Calendar.
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry, for the duration of study participation, and following completion of therapy for 5 months if female and 7 months if male.
* Female subjects of child-bearing potential must have a negative serum pregnancy test within 72 hours prior to receiving the first dose of study drug. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria: Has not undergone a hysterectomy or bilateral oophorectomy; or has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).

Exclusion Criteria

* Patients may not be receiving any other investigational agents. If received as part of first line treatment, last administration of previous investigational agent must be greater than 4 weeks prior to administration of study drug combination.
* Patients must not be pregnant or nursing due to the potential for congenital abnormalities or harm to nursing infants.
* Tumor harbors an epidermal growth factor receptor (EGFR) sensitizing (activating) mutation or an anaplastic lymphoma kinase (ALK) translocation. All other co-mutations will be allowed.
* Has known untreated central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are without evidence of progression for at least 4 weeks by repeat radiological imaging, clinically stable, and without requirement of steroid treatment for at least 14 days prior to first dose of study drug.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. Patients on chronic steroids (more than 4 weeks at stable dose) equivalent to ≤ 10mg prednisone will not be excluded.
* Has active autoimmune disease that has required systemic treatment in the past 1 year (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is acceptable.
* Has a known additional malignancy that is progressing and/or required active treatment within the past 3 years. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical or anal cancer, prostate cancer on stable dose of hormonal therapy without rising prostate-specific antigen (PSA), and breast cancer whom have been treated with curative intent, who may be on hormonal therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator.
* HIV positive with detectable viral load, or anyone not on stable anti-viral (HAART) regimen, or with <350 cluster of differentiation 4 (CD4+) T cells/microliter in the peripheral blood. No HIV testing is required.
* History of allogeneic hematopoietic cell transplantation or solid organ transplantation.
* Receipt of a live vaccine within 30 days of planned start of study medication
* History of interstitial lung disease (e.g., idiopathic pulmonary fibrosis, organizing pneumonia) or active, noninfectious pneumonitis that required immunosuppressive doses of glucocorticoids to assist with management. A history of radiation pneumonitis in the radiation field is permitted.
* Prisoners or subjects who are involuntarily incarcerated.
* Subjects who are compulsorily detained for treatment of either psychiatric or physical (e.g. infectious disease) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Maximal Tolerated Dose (MTD) | DLTs will be evaluated at the end of Cycle 1 (each cycle is 28 days)
  MTD is defined as the highest dose for which at most 1 patient out of 6 experiences a dose-limiting toxicity (DLT)
Overall Response Rate (ORR) | 2 years
  ORR is defined as achieving an objective response of either complete response or partial response

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 2 years
  Phase 2: PFS is defined as the duration of time from start of treatment to the first occurrence of disease progression or death on study from any cause, whichever occurs earlier.
Overall Survival (OS) at MTD | 2 years
  Phase 2: OS at MTD is defined as the time from the first dose of study treatment to the date of death (whatever the cause).

CONTACTS AND LOCATIONS:
Overall Officials: Rajwanth Veluswamy, MD, MSCR, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal.To achieve aims in the approved proposal.Proposals should be directed to xxx@yyy. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website (Link to be included).